CLINICAL TRIAL: NCT01220388
Title: Pilot Study of the Action L-lysine on Aldosterone and Cortisol Secretion in Healthy Volunteers.
Brief Title: Effects of L-lysine on Adrenal Secretion
Acronym: L-Lysine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple
Other Study IDs: 2008/138/HP
Record Dates: First submitted 2010-10-11; First posted 2010-10-13 (Estimated); Last update posted 2013-06-18 (Estimated); Status verified 2013-06

CONDITIONS: Male; Healthy Volunteers
Keywords: Aldosterone; L-lysine; Cortisol; Adrenal glands
MeSH Terms: interventions — Lysine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- L-lysine (Experimental): 11 days treatment with study drug, order of periods (active treatment or placebo) being sorted out.
  Interventions: Dietary Supplement: L-lysine
- placebo (Placebo Comparator): 11 days treatment with study drug, order of periods (L-lysine or placebo) being sorted out.
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: L-lysine — L-lysine, 4,95 G at day : 0,55 G 3 times a day, orally, during meals
  Arms: L-lysine
Dietary Supplement: placebo — placebo, 3 times a day, orally, during meals
  Arms: placebo

SUMMARY:
Data from the literature and previous in vitro research conducted in the investigators' laboratory (INSERM U413/EA4310, University of Rouen) suggest that adrenal corticosteroid secretion might be controlled by a paracrine mechanism involving serotonin type IV receptor (5-HT 4). L-lysine, a common amino-acid has been shown to act as a 5-HT4 agonist in vitro as well as in vivo. In the present physiology trial, plasma aldosterone and cortisol levels will be measured under treatment with aprepitant versus placebo, in both basal conditions and after activation of the adrenocortical function by various stimuli, including upright posture, metoclopramide, and after a 3 days salt-free diet. All healthy volunteers will be given two substances (L-lysine and placebo) in a random order during two 13 days periods separated by a 14 day-wash-out. This study should allow to determine the role of 5-HT4 receptors in the control of corticosteroid production in normal man.

DETAILED DESCRIPTION:
STUDY DESIGN Proof of concept, interventional, monocentric, randomised, double blind, cross-over study: The effects of L-lysine on corticosteroid secretion will be compared to those of a placebo. STUDY OBJECTIVES Main objective: to verify that adrenal corticosteroid secretion is actually controlled by L-lysine. Secondary objective: to determine the physiological conditions that involve the control of adrenocortical function by t5-HT4 receptors. NUMBER OF SUBJECTS 20 healthy volunteers ELIGIBILITY CRITERIA (see below) DURATION OF STUDY Overall duration: 13 months Inclusion period: 12 months Follow up period (for 1 subject): 5 weeks Exclusion period: 1 month ENDPOINTS PRIMARY ENDPOINT: blood aldosterone variation during orthostatic test SECONDARY ENDPOINTS Basal aldosterone alteration Aldosterone variation during metoclopramide & salt-free diet tests Basal and stimulated (3 different tests) alterations of renin, cortisol & ACTH REGULATORY AUTHORIZATIONS Ethics committee authorization: jan 21,2010 Regulatory authorization: july 9th 2010

ELIGIBILITY:
Inclusion Criteria:

* Male subjects;
* Age ranging 18 - 45 years old;
* Submitted to a social security regimen;
* Agreeing to the study & Informed consent form signed;
* Body mass index ([weight (kg)/height (m)]²) < 27;
* No treatment received 6 weeks before inclusion;
* No anomaly after: complete clinical examination, pulse measurement, ECG;
* Blood pressure on AMBP : Mean systolic blood pressure < 135 mmHg & Mean diastolic blood pressure < 85 mmHg
* No biological abnormality after biological testing o No participation in a clinical trial 3 months before inclusion.

Exclusion Criteria:

* Subject not agreeing to the study or impossible to follow-up;
* Known history of significant medical or surgical pathology, notably endocrine;
* Renal or hepatic insufficiency;
* Nephrotic syndrome;
* Edematous syndrome;
* Hypertension or postural hypotension;
* Cardiac rhythm or conduction pathologies;
* Cardiac insufficiency;
* Epilepsy;
* Significant psychiatric disorder;
* Known history of severe allergy, hypersensitivity to metoclopramide;
* Hereditary problems of fructose intolerance, glucose-galactose malabsorption or sucrase-isomaltase deficit;
* Impaired lactose tolerance.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2010-10; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Plasma aldosterone variation during orthostatic test | Day 5 of treatment, at each period

SECONDARY OUTCOMES:
Basal aldosterone alteration; Aldosterone variation during metoclopramide & salt-free diet tests; Basal and stimulated (3 different tests) alterations of renin, cortisol & ACTH | Day 5, 6, 7 and 11 of treatment, at each period

CONTACTS AND LOCATIONS:
Overall Officials: Hervé Lefebvre, PHD, Principal Investigator — University Hospital, Rouen
Locations (1):
- Rouen Clinical research Centre (CIC 0204), Rouen, France